CLINICAL TRIAL: NCT01167439
Title: Dysphagia in Oculopharyngeal Muscular Dystrophy. Evaluation, Endoscopic Examination of Swallowing, Treatment and Long Term Follow up.
Brief Title: Dysphagia in Oculopharyngeal Muscular Dystrophy (OPMD)- Evaluation, Endoscopic Examination of Swallowing, Treatment and Long Term Follow up
Acronym: OPMD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Itzhak Bravermen, MD, Hillel Yaffe Medical Center, Hadera, Israel
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0027-09-HYMC
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2009-12

CONDITIONS: Dysphagia
Keywords: OPMD, dysphagia; Dysphagia severity; Nutritional state; Speech quality; Upper esophageal sphincter myotomy
MeSH Terms: conditions — Deglutition Disorders; Muscular Dystrophy, Oculopharyngeal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mild dysphagia (No Intervention)
- Severe dysphagia (Active Comparator)
  Interventions: Procedure: Upper esophageal sphincter myotomy

INTERVENTIONS:
Procedure: Upper esophageal sphincter myotomy — Upper esophageal sphincter release operation to allow better swallowing. The intervention is done under GA and by extra-mucosal approach.
  Arms: Severe dysphagia

SUMMARY:
The investigators aimed to review the natural history of dysphagia and dysphonia in OPMD in order to identify the best candidates and the proper timing to perform dysphagia alleviating procedures in both heterozygote and homozygote patients from the large pool of cases with this disease in Israel.

DETAILED DESCRIPTION:
Clinical evaluation of patients suspected of having OPMD. Genetic confirmatory tests (diagnostic DNA test) at the genetic unit in Afula Hospital. Clinical follow-up with endoscopic fiber optic evaluation of swallowing. Pre-operative assessment. Crycopharyngeal myotomy intervention in selected patients. Nutrition follow-up.

ELIGIBILITY:
Inclusion Criteria:

* heterozygote and homozygote OPMD patients

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Dysphagia, quality of life. Proper intervention timing in OPMD based on knowledge about the natural history of the feeding difficulty. | at least 3 years
  Dysphagia, quality of life. Proper intervention timing in OPMD patients is very important and must be based on deep knowledge about the natural history of the feeding difficulty.

CONTACTS AND LOCATIONS:
Locations (1):
- Israel National Center for OPMD and Dysphagia, HYMC, POB 169, Hadera, Israel